CLINICAL TRIAL: NCT01503476
Title: RD-40 Development of Applications of the Bravo® pH Monitoring System and Evaluation of Its Performance
Brief Title: Development of Applications of the Bravo® pH Monitoring System and Evaluation of Its Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD-40
Record Dates: First submitted 2011-12-25; First posted 2012-01-04 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2015-07

CONDITIONS: Gastro Esophageal Reflux Disease
Keywords: gastro esophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esophageal pH Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental): healthy volunteers
  Interventions: Device: Bravo® pH Monitoring System
- symptomatic patients (Experimental): symptomatic patients with known or suspected gastro esophageal reflux disease
  Interventions: Device: Bravo® pH Monitoring System

INTERVENTIONS:
Device: Bravo® pH Monitoring System — Bravo pH monitoring
  Other Names: pH monitoring
  Arms: symptomatic patients
Device: Bravo® pH Monitoring System — Bravo pH monitoring
  Other Names: pH monitoring
  Arms: Healthy volunteers

SUMMARY:
Study Hypothesis:

This study is designed as an integral part of the development of new or improved features or components of the Bravo® pH Monitoring System and may serve verification and validation purposes The study population will include a group of healthy volunteers (Group A) and a group of symptomatic patients with known or suspected gastroesophageal reflux disease (Group B).

Group A: Healthy volunteers will not undergo invasive procedure. These volunteers may be asked to carry the capsule and\or Bravo Recorder. These procedures will serve to evaluate different technical matters such as human interface, ergonomic aspects and communication performances of the system Group B: Symptomatic patients will undergo invasive procedure, including Bravo capsule delivery, positioning and attachment. Confirmation of capsule attachment may be done by endoscopically.

These procedures will serve to evaluate overall system performance in actual clinical setup, for instance: Bravo Recorder performance including communication quality, human interface and similar, ergonomics of delivery device, pH Capsule performance, etc.

Subjects from both study groups as well as physician may be asked to provide feedback on the procedure and/or document their activities during the procedure.

DETAILED DESCRIPTION:
Up to a total of 220 subjects will participate in this study. The study will include two separate population groups. Group A of up to 170 healthy volunteers and Group B of up to 50 symptomatic patients with known or suspected gastro esophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 years old
2. Subject received an explanation about the nature of the study and agrees to provide written informed consent.

   Group A (healthy volunteers) Only
3. Subject is an healthy volunteer

Group B (symptomatic patients) Only 1. The subject was referred for pH monitoring procedure to detect acid reflux for at least one of the following reasons:

* Burning substernal chest pain (heartburn)
* Regurgitation of food or stomach contents
* Dysphagia
* Epigastric pain
* Non-erosive reflux disease (NERD)

Exclusion Criteria:

Group A and B-

1. Subject has a cardiac pacemaker or other implanted electromedical device.
2. Subject has any condition, which precludes compliance with study and/or device instructions.
3. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
4. Subject suffers from life threatening conditions
5. Subject currently participating in another clinical study which may interfere with study objectives, per physician discretion

   Additional exclusion criteria for Group B only
6. Subject has prior abdominal surgery other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
7. Subject is schedule to undergo MRI examination within 30 days from pH monitoring procedure.
8. Subject has known bleeding diathesis, strictures, severe esophagitis, varices and or obstructions -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of data samples transmitted by the capsule and successfully received by the receiver (e.g. percent of missed samples and percent of corrupted samples) | up to 96 hours
  Percentage of data samples in healthy volunteers and patients transmitted by capsule and successfully received by the receiver (e.g. percent of missed samples and percent of corrupted samples)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Adler, M.D., Principal Investigator — Bikur Holim medical center
Locations (1):
- Bikur Holim medical center, Jerusalem, Israel